CLINICAL TRIAL: NCT00944853
Title: The Effect of Zinc Supplementation, Provided as Either a Liquid Zinc Solution or Dispersible Tablets, on Plasma Zinc Concentration Among Young Burkinabe Children
Brief Title: Effects of Liquid Zinc Supplementation and Dispersible Zinc Tablets on Plasma Zinc Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Université Polytechnique de Bobo-Dioulasso (Other); Helen Keller International (Other); Nutriset (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 200917272; ZincTab
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2010-02

CONDITIONS: Zinc Deficiency
Keywords: zinc supplement; prevention; zinc deficiency; plasma zinc concentration
MeSH Terms: interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Zinc syrup (Experimental): Liquid Zinc Syrup (ZnSO4) solution provided daily
  Interventions: Dietary Supplement: Liquid zinc syrup
- Zinc tablet (Experimental): Dispersible zinc tablets provided daily
  Interventions: Dietary Supplement: Zinc tablet
- Placebo (Placebo Comparator): Liquid placebo supplement provided daily
  Interventions: Dietary Supplement: Liquid placebo supplement

INTERVENTIONS:
Dietary Supplement: Liquid zinc syrup — Liquid zinc syrup containing 5 mg zinc as zinc sulfate
  Other Names: Phytofla, Banfora, Burkina Faso
  Arms: Zinc syrup
Dietary Supplement: Zinc tablet — Dispersible zinc tablet containing 5 mg zinc
  Other Names: Nutriset S.A.S., France
  Arms: Zinc tablet
Dietary Supplement: Liquid placebo supplement — Liquid placebo supplement containing 0 mg zinc
  Other Names: Phytofla, Banfora, Burkina Faso
  Arms: Placebo

SUMMARY:
The study aims to compare the effects of two different formulations of zinc supplements on plasma zinc concentrations among young Burkinabe children.

DETAILED DESCRIPTION:
1) To investigate the effects of short-term zinc supplementation, provided either as a dispersible tablet containing zinc sulfate ("ZinCfant," Nutriset Ltd; Malaunay, France) or as a liquid ZnSO4 solution, on changes in serum zinc concentration, compared with a placebo in young Burkinabe children; and 2) to assess the relationship between change in serum zinc concentration and the presence of altered intestinal permeability within each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* currently breast feeding
* informed consent of a parent or guardian.

Exclusion Criteria:

* symptomatic acute or chronic febrile infections
* diarrhea within the past week
* consuming vitamin or mineral supplements or zinc-fortified infant formulas

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 462 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma zinc concentration | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Brown, MD, Principal Investigator — University of California, Davis
Locations (1):
- Toussiana Health District, Touziana, Burkina Faso

REFERENCES:
- [Result] Wessells KR, Ouedraogo ZP, Rouamba N, Hess SY, Ouedraogo JB, Brown KH. Short-term zinc supplementation with dispersible tablets or zinc sulfate solution yields similar positive effects on plasma zinc concentration of young children in Burkina Faso: a randomized controlled trial. J Pediatr. 2012 Jan;160(1):129-35.e3. doi: 10.1016/j.jpeds.2011.06.051. Epub 2011 Aug 25. PMID 21871635
- [Derived] Wessells KR, Peerson JM, Brown KH. Within-individual differences in plasma ferritin, retinol-binding protein, and zinc concentrations in relation to inflammation observed during a short-term longitudinal study are similar to between-individual differences observed cross-sectionally. Am J Clin Nutr. 2019 May 1;109(5):1484-1492. doi: 10.1093/ajcn/nqz014. PMID 30976780
- [Derived] Wessells KR, Hess SY, Ouedraogo ZP, Rouamba N, Ouedraogo JB, Brown KH. Asymptomatic malaria infection affects the interpretation of biomarkers of iron and vitamin A status, even after adjusting for systemic inflammation, but does not affect plasma zinc concentrations among young children in Burkina Faso. J Nutr. 2014 Dec;144(12):2050-8. doi: 10.3945/jn.114.200345. Epub 2014 Oct 1. PMID 25411038
- [Derived] Wessells KR, Hess SY, Rouamba N, Ouedraogo ZP, Kellogg M, Goto R, Duggan C, Ouedraogo JB, Brown KH. Associations between intestinal mucosal function and changes in plasma zinc concentration following zinc supplementation. J Pediatr Gastroenterol Nutr. 2013 Sep;57(3):348-55. doi: 10.1097/MPG.0b013e31829b4e9e. PMID 23689263